CLINICAL TRIAL: NCT04192799
Title: Comparative Effectiveness of Direct Admission & Admission Through Emergency Departments for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Nationwide Children's Hospital (Other); Providence Health & Services (Other); University of Pittsburgh (Other); Dartmouth College (Other); Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, JoAnna K. Leyenaar, Vice Chair of Research and Associate Professor, Department of Pediatrics, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IHS-2018C2-12902-IC
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-08

CONDITIONS: Hospitalization; Child Health

STUDY DESIGN:
Intervention Model Description: stepped-wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Admission (Experimental): Referring providers contact the hospital to arrange for a child to be admitted directly into the pediatric hospital medicine unit.
  Interventions: Behavioral: Direct admission
- ED Admission (Active Comparator): Children initially present at the Emergency Department and are then admitted to the pediatric hospital medicine unit.
  Interventions: Behavioral: ED admission

INTERVENTIONS:
Behavioral: Direct admission — Process of pediatric admission is through admission directly into the pediatric hospital medicine unit
  Arms: Direct Admission
Behavioral: ED admission — Process of pediatric admission is through the emergency department
  Arms: ED Admission

SUMMARY:
At a national level, emergency departments (EDs) serve as the portal of hospital admission for 75% of hospitalized children. The remainder occur via direct admission, defined as admission to hospital without first receiving care in the hospital's ED. The overall goals of this research are to: (i) implement pediatric direct admission systems at 3 hospitals, (ii) compare the timeliness of healthcare delivery for children who are admitted directly and through emergency departments, (iii) determine which patient populations achieve the greatest benefits from direct admission, and (iv) identify barriers and facilitators of successful implementation.

DETAILED DESCRIPTION:
The Specific Aims of this research are to: (i) Determine the effect of a pediatric direct admission system on timeliness of healthcare provision (the investigator's primary outcome), family experience of care, and rates of clinical deterioration compared to hospital admission beginning in the ED; (ii) Identify the pediatric populations and conditions that experience the greatest benefits from direct admission; and (iii) Through interviews with key informants, identify barriers to and facilitators of implementing standardized direct admission processes.

To achieve these Aims, a stepped-wedge cluster randomized controlled trial at three geographically diverse hospitals in the United States will be conducted, randomizing primary and urgent care practices in the hospitals' catchment area to cross over to the direct admission intervention at four time points. Linear models with random effects for clusters and time period fixed effects will be used to evaluate outcomes associated with the direct admission intervention. To examine for heterogeneity of treatment effects, interactions between direct admission and a priori-specified subgroups will be examined.

ELIGIBILITY:
Inclusion Criteria

Child has one of the following presenting diagnoses:

* gastroenteritis
* dehydration
* skin and soft tissue infection
* urinary tract infection/pyelonephritis
* pneumonia
* viral infection not otherwise specified
* influenza

Exclusion Criteria

Ineligible children include those:

* with planned admissions (i.e., chemotherapy)
* admitted to non-pediatric hospital medicine services (i.e., intensive care)
* transferred from other hospitals

Ages: 30 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1997 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnna K Leyenaar, MD, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Geisel School of Medicine at Dartmouth
Locations (3):
- United States (3):
  - Nationwide Children's Hospital, Columbus, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Providence Regional Medical Center - Everett, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leyenaar JK, McDaniel CE, Acquilano SC, Schaefer AP, Bruce ML, O'Malley AJ. Comparative effectiveness of direct admission and admission through emergency departments for children: a randomized stepped wedge study protocol. Trials. 2020 Nov 30;21(1):988. doi: 10.1186/s13063-020-04889-9. PMID 33256850

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinical practices
Groups:
- Sequence 1: Periods 1-4 With Direct Admission Intervention: Intervention: clinical practices received training in direct admissions for patients.
  Referring providers contact the hospital to arrange for a child to be admitted directly into the pediatric hospital medicine unit.
  Direct admission: Process of pediatric admission is through admission directly into the pediatric hospital medicine unit
- Sequence 2: Periods 2-4 With Direct Admission Intervention; Sequence 3: Periods 3-4 With Direct Admission Intervention; Sequence 4: Period 4 With Direct Admission Intervention: Intervention: clinical practices received training in direct admissions for patients.
  Referring providers contact the hospital to arrange for a child to be admitted directly into the pediatric hospital medicine unit.
  Direct admission: Process of pediatric admission is through admission directly into the pediatric hospital medicine unit
  ED admission: Process of pediatric admission is through the emergency department
Period: Step 1: Months 1-6
Arm/Group | Sequence 1: Periods 1-4 With Direct Admission Intervention | Sequence 2: Periods 2-4 With Direct Admission Intervention | Sequence 3: Periods 3-4 With Direct Admission Intervention | Sequence 4: Period 4 With Direct Admission Intervention
Started | 134; 18 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Patient Directly Admitted | 8; 18 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Patient Admitted Through ED | 126; 18 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Completed | 134; 18 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Not Completed | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Period: Step 2: Months 7-12
Arm/Group | Sequence 1: Periods 1-4 With Direct Admission Intervention | Sequence 2: Periods 2-4 With Direct Admission Intervention | Sequence 3: Periods 3-4 With Direct Admission Intervention | Sequence 4: Period 4 With Direct Admission Intervention
Started | 98; 18 Clinical practices | 60; 17 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Patient Directly Admitted | 8; 18 Clinical practices | 3; 17 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Patient Admitted Through ED | 90; 18 Clinical practices | 57; 17 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Completed | 98; 18 Clinical practices | 60; 17 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Not Completed | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Period: Step 3: Months 13-21
Arm/Group | Sequence 1: Periods 1-4 With Direct Admission Intervention | Sequence 2: Periods 2-4 With Direct Admission Intervention | Sequence 3: Periods 3-4 With Direct Admission Intervention | Sequence 4: Period 4 With Direct Admission Intervention
Started | 239; 18 Clinical practices | 146; 17 Clinical practices | 164; 17 Clinical practices | 0; 0 Clinical practices
Patient Directly Admitted | 23; 18 Clinical practices | 13; 17 Clinical practices | 9; 17 Clinical practices | 0; 0 Clinical practices
Patient Admitted Through ED | 216; 18 Clinical practices | 133; 17 Clinical practices | 155; 17 Clinical practices | 0; 0 Clinical practices
Completed | 239; 18 Clinical practices | 146; 17 Clinical practices | 164; 17 Clinical practices | 0; 0 Clinical practices
Not Completed | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices
Period: Step 4: Months 22-39
Arm/Group | Sequence 1: Periods 1-4 With Direct Admission Intervention | Sequence 2: Periods 2-4 With Direct Admission Intervention | Sequence 3: Periods 3-4 With Direct Admission Intervention | Sequence 4: Period 4 With Direct Admission Intervention
Started | 344; 18 Clinical practices | 246; 17 Clinical practices | 259; 17 Clinical practices | 307; 17 Clinical practices
Patient Directly Admitted | 28; 18 Clinical practices | 17; 17 Clinical practices | 18; 17 Clinical practices | 18; 17 Clinical practices
Patient Admitted Through ED | 316; 18 Clinical practices | 229; 17 Clinical practices | 241; 17 Clinical practices | 289; 17 Clinical practices
Completed | 344; 18 Clinical practices | 246; 17 Clinical practices | 259; 17 Clinical practices | 307; 17 Clinical practices
Not Completed | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices | 0; 0 Clinical practices

BASELINE CHARACTERISTICS:
Population: The above numbers reflect admissions that occurred following each clinic's respective DA program start date and which were included in the patient-level analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Admission | ED Admission | Total
Number analyzed (Participants) | 145 | 1852 | 1997
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2.8 [0.9 to 5.7] | 2.8 [1.1 to 6.9] | 2.8 [1.1 to 6.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 929 | 994
  Male | 80 | 923 | 1003
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 154 | 162
  Not Hispanic or Latino | 137 | 1645 | 1782
  Unknown or Not Reported | 0 | 53 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 10 | 130 | 140
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 670 | 699
  White | 93 | 819 | 912
  More than one race | 8 | 110 | 118
  Unknown or Not Reported | 4 | 120 | 124
Region of Enrollment [Number; unit: participants]
  United States | 145 | 1852 | 1997
Primary Payor [Count of Participants; unit: Participants] — Type of insurance
  Participants
    Medicaid | 68 | 1256 | 1324
    Commercial | 72 | 564 | 636
    Other | 5 | 32 | 37

OUTCOME MEASURES:

1. Primary Outcome: Timeliness of Clinical Care - Initial Therapeutic Management
Description: Length of time from arrival at the hospital until time of first antibiotics, IV placement, fluid administration, or other medications
Time Frame: within 6 hours of hospital admission
Population: These analyses include only those admissions that occurred following each clinic's respective DA program start date and for whom data were obtained.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Direct Admission | ED Admission
Number analyzed (Participants) | 139 | 1786
minutes | 142 [96.5 to 209.5] | 153 [85 to 258]
Statistical Analysis 1: Comparison: Direct Admission vs ED Admission; Test type: Equivalence — Testing was two-sided and p-values <0.05 were considered statistically significant; p < 0.001, Gamma Regression with Log Link Function — Testing was two-sided and p-values <0.05 were considered statistically significant, not adjusted for multiple comparison; Adjusted for demographics, clinical characteristics, time period; interaction term for hospital and time period, random effect for practice group; Mean Ratio = 0.74, 95% CI 2-sided [0.65 to 0.85]

2. Primary Outcome: Timeliness of Clinical Care - Initial Clinical Assessment
Description: Length of time from arrival at the hospital until first time when at least 3 vital signs were documented; if missing, time of initial brief nursing assessment
Time Frame: within 6 hours of hospital admission
Population: These analyses include all admissions that occurred following each clinic's respective DA program start date.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Direct Admission | ED Admission
Number analyzed (Participants) | 145 | 1852
minutes | 25 [19 to 31] | 13 [7 to 30]
Statistical Analysis 1: Comparison: Direct Admission vs ED Admission; Test type: Equivalence — Testing was two-sided and p-values <0.05 were considered statistically significant; p < 0.001, Gamma Regression with Log Link Function — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Ratio = 1.12, 95% CI 2-sided [1.06 to 1.19]

3. Primary Outcome: Timeliness of Clinical Care - Initial Diagnostic Testing
Description: Length of time from arrival at the hospital until time of initial labs and/or imaging, including "standing orders" for diagnostic testing in emergency departments
Time Frame: within 6 hours of hospital admission
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Direct Admission | ED Admission
Number analyzed (Participants) | 141 | 1,805
minutes | 120.5 [83 to 171] | 99 [48 to 186]
Statistical Analysis 1: Comparison: Direct Admission vs ED Admission; Test type: Equivalence — Testing was two-sided and p-values <0.05 were considered statistically significant; p = 0.37, Gamma Regression with Log Link Function — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Ratio = 0.93, 95% CI 2-sided [0.80 to 1.09]

4. Secondary Outcome: Number of Participants With Clinical Deterioration
Description: Transfer for pediatric intensive care or rapid response calls
Time Frame: within 6 hours of arrival on the inpatient unit
Population: These analyses include 145 DAs and 1852 ED admissions that occurred following each clinic's respective DA program start date.
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Admission | ED Admission
Number analyzed (Participants) | 145 | 1852
Participants | 1 | 15
Statistical Analysis 1: Comparison: Direct Admission vs ED Admission; Test type: Equivalence — Testing was two-sided and p-values <0.05 were considered statistically significant; p = 0.81, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.14 to 12.27]

5. Secondary Outcome: Pediatric Hospitalization Admission Survey of Experience (PHASE)
Description: Standardized closed-ended survey questions regarding parent-reported experience of hospital admission with respect to the admission process, communication with families, communication between providers, and the hospital space; composite measure on 0-1 scale, with higher scores indicating better family experience
Time Frame: Within 72 hours of hospital admission
Population: As a secondary, self-reported outcome measure, we only obtained data from the subsample of families who completed a PHASE survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Direct Admission | ED Admission
Number analyzed (Participants) | 67 | 805
score on a scale | 0.75 (0.22) | 0.71 (0.22)
Statistical Analysis 1: Comparison: Direct Admission vs ED Admission; Test type: Equivalence — Testing was two-sided and p-values <0.05 were considered statistically significant; p = 0.12, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Slope = 0.05, 95% CI 2-sided [-0.01 to 0.11]

ADVERSE EVENTS:
Time Frame: 6 hours (first 6 hours post inpatient admission)
Description: This study was deemed minimal risk by the IRB and reviewed as an expedited study. We did not expect any mortality or serious adverse events; possible adverse events included discomfort with completing the survey and loss of confidentiality.
Arm/Group | Direct Admission | ED Admission
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/1852
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/1852
Other Adverse Events (participants affected / at risk) | 0/145 | 0/1852
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Direct Admission (N=145) | ED Admission (N=1852)
(General disorders) | 0 (0) | 0 (0) — No SAEs expected

LIMITATIONS AND CAVEATS:
This study was implemented six weeks prior to the COVID-19 pandemic, which led to unprecedented changes to healthcare. Early in the pandemic, closures of primary care clinics, transitions to telehealth, and low ED volumes may have decreased DA access and improved relative timeliness of ED care. Throughout the study, pandemic-associated staffing challenges, shortages of bed availability, and pediatric unit closures (which were observed nationally) continued to impact the project.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT04192799/Prot_SAP_000.pdf